CLINICAL TRIAL: NCT04515576
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple-Ascending Subcutaneous Doses of LY3493269 in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of LY3493269 in Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17530; J1X-MC-GZHC (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-08-14; First posted 2020-08-17 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 1.5 milligrams (mg) Dulaglutide (Active Comparator): Participants received 1.5 mg dulaglutide subcutaneously (SC) once weekly (QW) for 4 weeks.
  Interventions: Drug: Dulaglutide
- 0.3 mg LY3493269 (Experimental): Participants received 4 fixed dosed of 0.3 mg LY3493269 SC QW for 4 weeks.
  Interventions: Drug: LY3493269
- 1 mg LY3493269 (Experimental): Participants received 4 fixed dosed of 1 mg LY3493269 SC QW for 4 weeks.
  Interventions: Drug: LY3493269
- 0.75/1.5/3 mg LY3493269 (Experimental): Participants received LY3493269 0.75 mg on week 1, 1.5 mg on week 2 and 3 mg on week 3 and 4 SC as weekly doses.
  Interventions: Drug: LY3493269
- 1.5/3/4/5 mg LY3493269 (Experimental): Participants received LY3493269 1.5 mg on week 1, 3 mg on week 2, 4 mg on week 3 and 5 mg on week 4 as weekly doses.
  Interventions: Drug: LY3493269
- Placebo (Placebo Comparator): Participants received placebo subcutaneously (SC) once weekly (QW) for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3493269 — Administered SC
  Arms: 0.3 mg LY3493269; 0.75/1.5/3 mg LY3493269; 1 mg LY3493269; 1.5/3/4/5 mg LY3493269
Drug: Dulaglutide — Administered SC
  Other Names: LY2189265
  Arms: 1.5 milligrams (mg) Dulaglutide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine the side effects related to LY3493269 in participants with type 2 diabetes. Blood tests will be performed to check concentrations of LY3493269 in the bloodstream. Each enrolled participant will receive LY3493269, dulaglutide, or placebo. The study will last up to approximately 16 weeks for each participant and may include up to 11 visits.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female not of childbearing potential
* Have a body mass index of 23 to 50 kilograms per square meter (kg/m²), inclusive, at screening
* Have had a stable body weight (<5% body weight change) for the 3 months prior to screening
* Have not modified their diet or adopted any nutritional lifestyle modification in the 3 months prior to screening
* Have type 2 diabetes mellitus (T2DM) controlled with diet and exercise alone or are on a stable dose of metformin for at least 3 months before screening. Patients with comorbid conditions commonly associated with diabetes (for example, hypertension, hypercholesterolemia, hypothyroidism) may be eligible for inclusion if conditions are assessed by the investigator to be well controlled and stable for at least 3 months prior to screening
* Have an HbA1c of at least 7.0% and no more than 10.5% at screening
* Have clinical laboratory test results within the normal range for the population or investigative site, or with abnormalities deemed not clinically significant by the investigator

Exclusion Criteria:

* Have type 1 diabetes mellitus or latent autoimmune diabetes in adults
* Have uncontrolled diabetes, defined as an episode of ketoacidosis or hyperosmolar state requiring hospitalization in the 6 months prior to screening
* Have a history of proliferative diabetic retinopathy, diabetic maculopathy, or severe nonproliferative diabetic retinopathy that requires acute treatment
* Have had more than 1 episode of severe hypoglycemia, as defined by the American Diabetes Association criteria, within 6 months before screening or has a history of hypoglycemia unawareness or poor recognition of hypoglycemic symptoms.
* Have a definitive diagnosis of autonomic neuropathy as evidenced by urinary retention, resting tachycardia, orthostatic hypotension, or diabetic diarrhea
* Have a history of acute or chronic pancreatitis
* Have a self or family history (first-degree relative) of multiple endocrine neoplasia type 2A or type 2B, thyroid C-cell hyperplasia, or medullary thyroid carcinoma
* Have calcitonin levels of 20 picograms per millilitre (pg/mL) or more at screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Miami Research Associates, Miami, Florida
  - Clinical Trials of Texas, Inc., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3493269 in Participants With Type 2 Diabetes — https://trials.lillytrialguide.com/en-US/trial/1xujziv0yfFVul40lqzrPv

RESULTS

PARTICIPANT FLOW:
Groups:
- 1.5 Milligrams (mg) Dulaglutide: Participants received 1.5 mg dulaglutide SC QW for 4 weeks.
Period: Overall Study
Arm/Group | Placebo | 1.5 Milligrams (mg) Dulaglutide | 0.3 mg LY3493269 | 1 mg LY3493269 | 0.75/1.5/3 mg LY3493269 | 1.5/3/4/5 mg LY3493269
Started | 7 | 8 | 8 | 8 | 11 | 14
Received at Least One Dose of Study Drug | 7 | 8 | 8 | 8 | 11 | 14
Completed | 7 | 8 | 8 | 8 | 11 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- 1.5 mg Dulaglutide: Participants received 1.5 mg dulaglutide SC QW for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | 1.5 mg Dulaglutide | 0.3 mg LY3493269 | 1 mg LY3493269 | 0.75/1.5/3 mg LY3493269 | 1.5/3/4/5 mg LY3493269 | Total
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 11 | 14 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (6.7) | 63.3 (6.6) | 60.9 (5.6) | 59.8 (3.4) | 55.1 (5.3) | 59.9 (6.9) | 59.2 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 4 | 6 | 6 | 25
  Male | 3 | 5 | 6 | 4 | 5 | 8 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 5 | 8 | 9 | 13 | 46
  Not Hispanic or Latino | 0 | 4 | 3 | 0 | 2 | 1 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 1 | 1 | 4
  White | 7 | 7 | 5 | 8 | 10 | 13 | 50
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 8 | 8 | 8 | 11 | 14 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Treatment-Emergent Adverse Event(s) (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: TEAE is an untoward medical occurrence that emerges during a defined treatment period, having been absent pretreatment, or worsens relative to the pretreatment state, and does not necessarily have to have a causal relationship with this treatment.
  An SAE is defined as any untoward medical occurrence that, at any dose:
  1. Results in death
  2. Is life-threatening
  3. Requires inpatient hospitalization or prolongation of existing hospitalization
  4. Results in persistent disability/incapacity
  5. Is a congenital anomaly/birth defect
  6. Other situations: Based on medical or scientific judgement.
  A summary of SAEs, TEAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module
Time Frame: Baseline through final follow-up at Day 57
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 1.5 mg Dulaglutide | 0.3 mg LY3493269 | 1 mg LY3493269 | 0.75/1.5/3 mg LY3493269 | 1.5/3/4/5 mg LY3493269
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 11 | 14
Participants
  SAEs Related to Study Drug Administration | 0 | 0 | 0 | 0 | 0 | 0
  TEAEs Related to Study Drug Administration | 2 | 5 | 3 | 7 | 10 | 13

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to 168 Hours Postdose AUC(0-168) of LY3493269
Description: Area Under the Concentration Versus Time Curve from Time Zero to 168 Hours Postdose AUC(0-168) of LY3493269
Time Frame: Predose, 6, 12, 24, 48, 72, 96 and 168 h postdose at Weeks 1 and 4.
Population: All participants who received at least one dose of LY3493269 and had evaluable PK data.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Groups:
- 0.3 mg LY3493269 QW: Participants received 4 fixed dosed of 0.3 mg LY3493269 SC QW for 4 weeks.
- 1 mg LY3493269 QW: Participants received 4 fixed dosed of 1 mg LY3493269 SC QW for 4 weeks.
- 0.75/1.5/3 mg LY3493269 QW: Participants received LY3493269 0.75 mg on week 1, 1.5 mg on week 2 and 3 mg on week 3 and 4 SC as weekly doses.
- 1.5/3/4/5 mg LY3493269 QW: Participants received LY3493269 1.5 mg on week 1, 3 mg on week 2, 4 mg on week 3 and 5 mg on week 4 as weekly doses.
Arm/Group | 0.3 mg LY3493269 QW | 1 mg LY3493269 QW | 0.75/1.5/3 mg LY3493269 QW | 1.5/3/4/5 mg LY3493269 QW
Number analyzed (Participants) | 8 | 8 | 11 | 11
nanogram*hour per milliliter (ng*h/mL)
  Week 1 | 4220 (27) | 18500 (40) | 10200 (30) | 22800 (25)
  Week 4: number analyzed (Participants) | 8 | 8 | 11 | 5
  Week 4 | 10600 (21) | 38500 (25) | 105000 (27) | 123000 (22)

3. Secondary Outcome: PK: Maximum Observed Drug Concentration (Cmax) of LY3493269
Description: Maximum Observed Drug Concentration (Cmax) of LY3493269
Time Frame: Predose, 6, 12, 24, 48, 72, 96 and 168 h postdose at Weeks 1 and 4.
Population: All participants who received at least one dose of LY3493269 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 0.3 mg LY3493269 QW | 1 mg LY3493269 QW | 0.75/1.5/3 mg LY3493269 QW | 1.5/3/4/5 mg LY3493269 QW
Number analyzed (Participants) | 8 | 8 | 11 | 14
nanogram per milliliter (ng/mL)
  Week 1 | 31.2 (31) | 153 (51) | 73.6 (32) | 165 (34)
  Week 4: number analyzed (Participants) | 8 | 8 | 11 | 5
  Week 4 | 80.3 (22) | 287 (26) | 818 (28) | 920 (28)

4. Secondary Outcome: Pharmacodynamics (PD):Change From Baseline to Day 29 in Fasting Plasma Glucose
Description: Pharmacodynamics (PD): Summary Statistics (Mean, Standard Deviation) of Change From Baseline to Day 29.
Time Frame: Baseline, Day 29
Population: All participants who received at least one dose of study drug and had evaluable fasting plasma glucose data.
Measure: Mean (Standard Deviation); unit: millimoles per litre (mmol/L)
Arm/Group | Placebo | 1.5 mg Dulaglutide | 0.3 mg LY3493269 | 1 mg LY3493269 | 0.75/1.5/3 mg LY3493269 | 1.5/3/4/5 mg LY3493269
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 11 | 13
millimoles per litre (mmol/L) | -1.07 (2.34) | -4.11 (2.82) | -2.20 (1.47) | -4.83 (2.75) | -3.61 (3.29) | -3.98 (3.11)

ADVERSE EVENTS:
Time Frame: Baseline through final follow-up at Day 57
Description: All participants who received at least one dose of study drug.
Groups:
- 1.5 mg Dulaglutide QW: Participants received 1.5 mg dulaglutide SC QW for 4 weeks.
Arm/Group | Placebo | 1.5 mg Dulaglutide QW | 0.3 mg LY3493269 QW | 1 mg LY3493269 QW | 0.75/1.5/3 mg LY3493269 QW | 1.5/3/4/5 mg LY3493269 QW
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/8 | 0/8 | 0/11 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/8 | 0/8 | 0/11 | 0/14
Other Adverse Events (participants affected / at risk) | 2/7 | 5/8 | 5/8 | 7/8 | 11/11 | 13/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=7) | 1.5 mg Dulaglutide QW (N=8) | 0.3 mg LY3493269 QW (N=8) | 1 mg LY3493269 QW (N=8) | 0.75/1.5/3 mg LY3493269 QW (N=11) | 1.5/3/4/5 mg LY3493269 QW (N=14)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 2 (2)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (8) | 2 (2) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (6) | 5 (5)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (15) | 3 (3) | 4 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 4 (6) | 3 (3) | 5 (9)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (9)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site dermatitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Tenderness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 5 (5) | 3 (4) | 8 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (6) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 7 (7) | 7 (8)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Withdrawal hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT04515576/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/76/NCT04515576/SAP_001.pdf